CLINICAL TRIAL: NCT03379519
Title: The Development and Evaluation of Multi-domain Attention Training for Older Adults With Mild Cognitive Impairment
Brief Title: Protocol of Multi-domain Attention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yang, Hui-Ling, Ph.D. candidate, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N201602069
Record Dates: First submitted 2017-12-10; First posted 2017-12-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-domain Attention Training (MAT) (Experimental): Training sessions of the MAT group is 45 minutes/day, 3 sessions/week, for 12 weeks (36 sessions).
  Interventions: Behavioral: Multi-domain Attention Training (MAT)
- Passive information activities (PIA) (Active Comparator): The training sessions of PIA is the same as MAT group (45 min/day, 3 days/week, for 12 weeks, for a total of 36 sessions).
  Interventions: Behavioral: Passive information activities (PIA)

INTERVENTIONS:
Behavioral: Multi-domain Attention Training (MAT) — The training content emphasis three concept of attention include: intensity of attention, executive attention, and spatial orienting attention.
  Other Names: Attention training
  Arms: Multi-domain Attention Training (MAT)
Behavioral: Passive information activities (PIA) — The active control group (Passive information activities) training content included reading online e-books and playing online games.
  Other Names: Active control group
  Arms: Passive information activities (PIA)

SUMMARY:
This study sought to investigate the changes in attention in older adults with mild cognitive impairment after Multi-domain Attention Training .

DETAILED DESCRIPTION:
This double-blind randomized controlled study has a 2-arm parallel group design. All subjects will be randomized by the block randomization, into intervention group (Multi-domain Attention Training, MAT), or active control group (Passive information activities, PIA). Training sessions of the MAT group are 45 minutes/day, 3 days/week, for 12 weeks (36 sessions each). The training of PIA group is the same as MAT group. The investigators constructed a rigorous MAT program adhering to the Consolidated Standards of Reporting Trials (CONSORT) reporting guidelines. The investigators expect to determine the improvement in attention function of older adults with mild cognitive impairment after using the MAT program.

ELIGIBILITY:
Inclusion Criteria:

* Participants must endorse at least two items from a list of frequent subjective memory complaints by patient and/or an informant
* Objective memory impairment on neuropsychological tests of memory 1.5 SD or more below age/education norms
* Clinical neurologic examination by the Mini-Mental State Examination (MMSE) score of 24 or higher
* No impairment in personal activities of daily living (P-ADL) as determined by clinical interview with participant and family

Exclusion Criteria:

* The clinical diagnosis of dementia was based on the DSM-IV-TR
* Active in another cognitive or memory-related training in the past year
* Comorbid medical conditions that would predispose them to imminent functional decline or cognitive impairment
* A diagnosis of major neurological or psychiatric illness history and/or behavioral problems that would sufficiently impair performance to make participation impossible
* Severe losses in vision, hearing, or communicative ability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in attention as measured by the Digit Span Task (DS). | Change from baseline in executive attention at Immediate post-test, 3 months, 6 months after intervention.
  The primary outcome indicators is executive attention assessed by the Digit Span Task (DS).

SECONDARY OUTCOMES:
Change in attention as measured by the Trail Making Test (TMT). | Change from baseline in spatial orienting attention at Immediate post-test, 3 months, 6 months after intervention.
  The secondary outcome indicator is spatial orienting attention evaluated by the Trail Making Test.

IPD SHARING:
Plan to Share IPD: No